CLINICAL TRIAL: NCT02409810
Title: Safety, Feasibility, and Acceptability of Patient-Controlled Anxiolysis With Dexmedetomidine (PCA-DEX) for Burn-care Dressing Changes
Brief Title: Patient-Controlled Anxiolysis With Dexmedetomidine (PCA-DEX) for Burn-care Dressing Changes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015H0019
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Results first posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Anxiety; Burns
MeSH Terms: conditions — Anxiety Disorders; Burns | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PCA-DEX Patients (Experimental): Prior to the burn dressing changes PCA-DEX patients will receive a bolus of dexmedetomidine (Precedex®) 0.25 mcg/kg administered over 10mins by nurse staff, followed by a continuous infusion of Precedex® at 0.4 mcg/kg/hr via a standard infusion pump (LifeCare PCA). Patients will self-medicate as needed for anxiety self-management by self-administering a bolus of Precedex® 0.1 mcg/kg.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Prior to the burn dressing changes PCA-DEX patients will receive a bolus of dexmedetomidine (Precedex®) 0.25 mcg/kg administered over 10 minutes by nursing staff, followed by a continuous infusion of Precedex® at 0.4 mcg/kg/hr via a standard infusion pump (LifeCare PCA). Patients will self-medicate as needed for anxiety self-management by self-administering a bolus of Precedex® 0.1 mcg/kg. This dosage is within the FDA-approved package insert parameters. Heart rate, blood pressure and oxygen saturation will be closely monitored by a staff RN already trained to provide care in the procedure room. 1 hour prior to- and after completion of the burn dressing change each day using a 100-mm visual analog scale. Patients will both rate their satisfaction with PCA-DEX for anxiety management after each completion of the burn dressing change.
  Other Names: Precedex, PCS-DEX

SUMMARY:
The primary aim of this pilot study is to establish the safety and feasibility of patient-controlled administration with dexmedetomidine for anxiolysis (PCA-DEX) during burn care dressings for patients with burn injury. The secondary aim is to determine the acceptability of PCA-DEX for anxiety symptom management by patients with burn injury and nursing staff caring for these patients. Objectives Primary Aim #1 Safety: To examine the safety of PCA-DEX as determined by the proportion of patients successfully completing the pilot trial without adverse effect which include significant hypotension, bradycardia, or agitation from uncontrolled anxiety. Primary Aim #2 Feasibility: The primary objective of this study is to establish feasibility of subject recruitment and protocol adherence in a pilot study of PCA-DEX in patients with burn injury requiring dressing changes. Feasibility will be defined by the following criteria: a) number and proportion of patients who consent to enrollment, b) proportion of eligible subjects enrolled prior to first dressing change, c) number of days on protocol that patients successfully use the PCS device, d) ability of burn nurses to adjust the pump and adhere to the infusion rates of the PCA-DEX protocol. Secondary Aim #1 Patient Acceptability: A secondary objective of this pilot study is to have patients evaluate PCA-DEX in regards to patients' willingness to use PCA-DEX prior to and during burn dressing changes to self-manage anxiety and their satisfaction ratings with anxiety self-management. Secondary Aim #2 Nurse Acceptability: Another secondary aim of this pilot study is to evaluate the nursing staffs' acceptability of the PCA-DEX protocol for patients' to self-manage anxiety surrounding burn care dressing changes. Hypotheses #1: PCA-DEX protocol will be safe to administer during burn care dressing changes. #2: PCA-DEX will be feasible to implement on the Burn Center at OSUWMC. #3: Patients will favorably appraise PCA-DEX for the self-control of anxiety associated with burn care dressing changes, and be satisfied with PCA-DEX for the management of anxiety. #4: Nursing Staff will favorably appraise PCA-DEX while performing burn care dressing changes.

DETAILED DESCRIPTION:
Study Procedures Dexmedetomidine PCA Protocol: The PCA-DEX dosing algorithm will consist of a loading dose (0.25 mcg/kg) given intravenously over 10 minutes, administered 10 minutes prior to the start of burn wound care, followed by a continuous basal infusion of 0.4 mcg/kg/hr with 6 allowable patient-controlled self-boluses per hour (0.1 mcg/kg) each with a 10-minute lock-out. Drs. Larry Jones and J. Kevin Bailey or their designate will write the PCA-DEX medication orders. Subjects will receive standard opioid therapy (oral oxycodone/acetaminophen 5/325 mg 60 min. prior and IV morphine 4-12 mg or hydromorphone IV 0.5-1.5 mg 5 to 10 min. prior and buccal fentanyl 400 mcg as needed during burn wound care) and can receive bolus supplemental sedative medications (benzodiazepines) as ordered by Drs. Jones or Bailey if needed in the judgment of the burn-care nurse. Subjects will be monitored closely by research personnel during the first burn wound care session from 1 hour prior to 1 hour after completion of burn wound care. Every heart rate and blood pressure recordings will be abstracted from the medical record from 1 hour prior to through 1 hour after completion of the daily burn wound dressing changes for days 1 through 5. Alert adverse events will be reported by research personnel or the patient-care nurse to first the attending physician and then to the safety monitor.

Nurse alert parameters to notify the attending physician and independent safety monitor include: heart rate (HR) < 55 beats per min sustained for > 10 min; systolic BP < 90 mm Hg or >140 mm Hg sustained for >10 minutes; diastolic BP < 50 mm Hg or >90 mm Hg sustained for >10 minutes, respiratory rate < 10 breaths per minute sustained for >10 minutes or oxygen saturation <92% sustained for >10 minutes; or persistent inability to understand rationale for triggering the PCA device despite education and demonstration.

If the study subject has evidence of sustained hemodynamic instability (HR<60 bpm, SBP <90 mmHg or DBP < 50 mmHg) during the daily pre-procedure assessment, the patient will not be eligible to receive study drug on that day. For that day the patient will receive standard of care as appropriate instead of the study intervention. The patient will then be reassessed prior to the subsequent study days to determine eligibility for study drug up through day 5.

Data Collection Measures and Procedures Study entry demographic and descriptive data: Data to be recorded includes: age, gender, race, ethnicity, admission weight, severity of burn injury, burn etiology, total body surface area burned and depth of injury, and all home and hospital medications.

Daily Measures on Protocol. The following will be obtained from enrolled patients each day by a member of the research team.

Overall anxiety and pain. The abbreviated Burn Specific Anxiety and Pain Scale (BSAPS) on day 1, 1 hour prior to the first burn dressing change.

Procedural Anxiety. Anxiety, defined as a state marked by apprehension, agitation, increased motor activity, arousal, and fearful withdrawal will be obtained from subjects. Patients will evaluate current anxiety level 1 hour before and 1 hour after each burn dressing change using a 100-mm Visual Analogue scale-anxiety (VAS-A). Subjects will be asked to rate their current level of anxiety on the VAS-A in response to, "How anxious are you feeling today?" A 100-millimeter vertical line will be anchored on each end by statements 'not anxious at all' to 'the most anxious I have ever been'. The VAS-A will have a vertical orientation, as it is more sensitive and easier for subjects to use, particularly for those with a narrowed visual field or when under stress. Subjects will be asked to mark their current anxiety level on the vertical line. Scores will be derived by the distance in millimeters from the bottom anchor to the mark placed by the subject, yielding interval level data. Reason(s) for not obtaining a daily anxiety assessment will be recorded. The proportion of those assessments completed and reasons for non-completion will be used to inform strategies to minimize missing data for our planned randomized clinical trial.

Procedural Pain. Patients' will evaluate current pain level 1 hour before and 1 hour after each burn dressing change using a 100-mm Visual Analogue Scale-Pain. Patients will be asked to rate their current level of pain on the VAS-P in response to "How much pain are you having right now?" A 100-millimeter vertical line will be anchored on each end by statements of 'no pain at all' to 'the most pain I have ever experienced'. As with the VAS-A, the vertical orientation has been chosen due to increased sensitivity and ease of use for patients.Subjects will be asked to mark their current pain level on the vertical line. Scores will be derived by the distance in millimeters from the bottom anchor to the mark placed by the subject, yielding interval level data. Reason(s) for not obtaining the pain assessments will be recorded. The proportion of those assessments completed and reasons for non-completion will be used to inform strategies to minimize missing data for our planned randomized clinical trial.

Protocol adherence. A checklist will be completed daily to monitor the number of days subjects are able to use the PCA device for up to 5 days. A checklist will also be used to monitor the ability of the burn-nurses to adhere to the PCA protocol per instructions.

Daily adverse event monitoring. Research staff will record and report the presence of hypotension, bradycardia (known adverse effects of dexmedetomidine), and protocol deviations related to drug, pump or both. Heart rate and blood pressure will be abstracted from the medical record. Research team staff or burn-nurses caring for PCA-DEX subjects will alert the attending physician and the safety monitor for HR < 55 bpm sustained for > 10 min; systolic BP < 90 mm Hg or >140 mm Hg sustained for >10 minutes; diastolic BP < 50 mm Hg or >90 mm Hg sustained for >10 minutes, respiratory rate < 10 breaths per minute sustained for >10 minutes or oxygen saturation <92% sustained for >10 minutes during the period 1 hour prior through 1 hour after completion of burn wound dressing change on days 1-5 for any necessary intervention or protocol withdrawal.

Post-PCA-DEX Acceptability Survey. Upon completion of the PCA-DEX protocol, we will query subjects and nurses about their satisfaction with self-administration of medication to manage anxiety, ease of medication administration, and the resulting level of relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18- 89 admitted for initial management of a thermal burn injury (flame, scald, contact) with >1% total body surface area
* Expected stay on the Burn Center for 3 or more days
* Read, write and speak English
* Burn injury experienced <48 hours prior to admission to the Burn Center for care

Exclusion Criteria:

* Patients who are pregnant
* Patients that are incarcerated
* Patients in active alcohol withdrawal
* Patients with current hemodynamic instability (current hypotension systolic blood pressure <100 mmHg, sustained heart rate < 60 beats/min without a pacemaker, symptomatic bradycardia, or second or third degree heart block)
* Cannot use push button PCA device (i.e., paralysis)
* Acute hepatitis
* Acute liver failure
* Acute stroke
* Acute seizures
* Acute myocardial infarction
* Severe cognition or communication difficulties (e.g., coma, deafness without signing literacy, dementia, non-English speaking)
* Chemical or electrical burn injury
* Any condition precluding inclusion at the discretion of the burn surgeons

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Jones, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCA-DEX Patients
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | PCA-DEX Patients
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 45.1 [45.1 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Successfully Completing the Pilot Trial Without Adverse Effects
Description: Post-PCA-DEX Acceptability Survey was completed to measure the Patient acceptability. Upon completion of the PCA-DEX protocol, subjects were asked about their satisfaction with self-administration of medication to manage anxiety, ease of medication administration, and the resulting level of relaxation by completing the PCA-DEX acceptability survey.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | PCA-DEX Patients
Number analyzed (Participants) | 20
Participants | 16

2. Primary Outcome: Feasibility Outcome #1 Number of Patients Who Consent to Enrollment
Description: Total patients who consented to enrollment among those in eligible patient population
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | PCA-DEX Patients
Number analyzed (Participants) | 20
Participants | 20

3. Primary Outcome: Feasibility Outcome #2 - Number of Patients Adhering to Protocol Over the Total Number of Eligible Intervention Days
Description: To establish feasibility by evaluating protocol adherence as defined by the total number of intervention days without protocol violation (defined as non-compliance with intervention implementation, infusion rates and/or pump adjustment) over the total number of eligible intervention days
Time Frame: 5 days
Measure: Number; unit: participants
Arm/Group | PCA-DEX Patients
Number analyzed (Participants) | 20
participants | 20

4. Secondary Outcome: Patient Acceptability (Number of Patients Willing to Use PCS-DEX Prior to and During Burn Dressing Changes)
Description: Patients evaluation of PCS-DEX in regards to their willingness to use PCA-DEX prior to and during burn dressing changes to self-manage anxiety and their satisfaction ratings with anxiety self-management.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | PCA-DEX Patients
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | PCA-DEX Patients
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT02409810/Prot_SAP_000.pdf